CLINICAL TRIAL: NCT03484780
Title: VisONE Pilot Study of Chronic Asymptomatic Diaphragmatic Stimulation for Patients With Symptomatic Heart Failure, Reduced Ejection Fraction and Preserved Ventricular Synchrony
Brief Title: VisONE Heart Failure Study: Pilot
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: VisCardia Inc. (Industry)
Collaborators: Clinical Accelerator (Industry); University of Glasgow (Other); University Hospital, Zürich (Other); Stiftung für Herz-und Kreislaufkrankheiten (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VisCardia H01_17
Record Dates: First submitted 2018-03-16; First posted 2018-04-02 (Actual); Last update posted 2020-05-20 (Actual); Status verified 2020-05

CONDITIONS: Heart Failure With Reduced Ejection Fraction, HFrEF
Keywords: Implantable Heart Failure Device Therapy; Asymptomatic Diaphragmatic Stimulation

STUDY DESIGN:
Intervention Model Description: Patients implanted with the VisONE implantable system for delivering chronic Asymptomatic Diaphragmatic Stimulation (ADS).
Masking Description: Independent data review and analysis by the University of Glasgow Department of Biostatistics
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- VisONE ADS (Experimental): Patients implanted with a VisONE stimulator and leads for receiving continual Synchronized Diaphragmatic Stimulation
  Interventions: Device: VisONE ADS

INTERVENTIONS:
Device: VisONE ADS — VisONE stimulator and leads for delivering continual Synchronized Diaphragmatic Stimulation
  Other Names: Synchronized Diaphragmatic Stimulation

SUMMARY:
The VisONE HF pilot is a feasibility pilot for evaluating the benefits and risks of chronically delivering Asymptomatic Diaphragmatic Stimulation in medical refractory heart failure patients using the VisONE™ implantable system for 12 months.

DETAILED DESCRIPTION:
This 12 month study is intended to validate the early benefits observed with Asymptomatic Diaphragmatic Stimulation (ADS) as a primary form of heart failure therapy with low rates and severity of adverse effects. Medical refractory symptomatic heart failure patients with reduced ejection fraction and no evidence of arrhythmias or ventricular dysynchrony will undergo laparoscopic implantation of the VisONE™ implantable system comprised of a pulse generator and two leads, programmed to deliver cardiac-gaited diaphragmatic stimulation pulses at asymptomatic outputs. Patients will be followed in pre-specified durations of 1,3,6 and 12-months using a series of evaluations of hemodynamic, echocardiographic, heart failure status, diaphragmatic function, implanted system data and standard safety measures including adverse events, for comparison with their baseline values. The results are intended to be used for designing a subsequent larger study for performing statistical power calculations.

ELIGIBILITY:
Inclusion Criteria

* NYHA class II/III medical refractory despite guideline indicated heart failure medications
* Sinus rhythm with <10% ectopy
* EF ≤ 35%
* NT-proBNP > 500 (250 if on loop diuretics)

Exclusion Criteria

* 6MHW >500 m or < 200 m
* Resting HR > 140 bpm
* SBP <80 mmHg or > 170 mmHg
* Serum creatine > 2.5 mg/dL
* Ventricular dyssynchrony by ECG with QRS ≥ 140ms
* Unstable angina, AMI, CABG, PTCA, CVA/TIA, persistent AF, NSVT, sustained VT or VF, or DCCV within 3 months
* Intermittent inotropic drug treatment
* Existing pacemaker or indications for a pacemaker
* Severe primary pulmonary disease including pulmonary arterial hypertension or severe COPD, or other respiratory or lung diseases where FEV < 50% or any condition with severe diaphragmatic dysfunction
* Previous open laparotomy within 1 year or contraindications to laparoscopy, as determined by implanting physician
* Known or active intra-abdominal infections, or known intra-abdominal pathology
* Previous thoracic or abdominal organ transplant, transplant waiting list
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2018-07-25 (Actual); Primary Completion 2019-12-12 (Actual); Study Completion 2019-12-12 (Actual)

PRIMARY OUTCOMES:
Freedom from serious complications or adverse events during procedural recovery and acute therapy | after 3 months of therapy
  The following serious complications and adverse events will be analyzed for their rate and severity and compared to other implantable device systems
  * Excessive procedural or implanted system morbidity
  * Procedural or implanted system events resulting in unscheduled patient hospitalizations and surgical intervention
  * Incidences resulting in physician choice to permanently discontinue therapy

SECONDARY OUTCOMES:
Freedom from complications or adverse events during chronic therapy | after 3 and 12 months of therapy
  The following adverse events will be analyzed for their rate and severity and compared to other implantable device systems
  * Procedural or implanted system events resulting in adverse patient symptoms
  * Degradation of respiratory function by spirometer measures associated with procedure or implanted system
  * Adverse events due to procedural or implanted system complications correctable by non re-operative means including system reprogramming or other readjustments
Freedom from serious complications or adverse events during chronic therapy | after 12 months of therapy
  The following serious complications and adverse events will be analyzed for their rate and severity and compared to other implantable device systems
  * Excessive procedural or implanted system morbidity
  * Procedural or implanted system events resulting in unscheduled patient hospitalizations and surgical intervention
  * Incidences resulting in physician choice to permanently discontinue therapy

OTHER OUTCOMES:
Clinical composite of heart failure and cardiac function | after 0, 1, 3, 6 and 12 months of therapy
  The following outcomes will be analyzed determine the potential therapeutic impact on clinical heart failure management
  * NT Pro-BNP blood levels to assess heart failure status
  * Improvements to cardiac output, stroke volume or left ventricular filling
  * Improvements to left ventricular volumes or ejection fraction
  * Improvements to heart failure status, 6 minute hall walk, or assessment by heart failure questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Vitaly Demyanchuk, M.D. Ph.D., Principal Investigator — Kyiv City Heart Center; Rudenko Vladimirovich, M.D., Principal Investigator — Amosov National Institute of Cardiovascular Surgery; Tamaz Shaburishvil, M.D., Principal Investigator — Tbilisi Heart and Vascular Clinic
Locations (3):
- Tbilisi Heart and Vascular Clinic, Tbilisi, Georgia
- Ukraine (2):
  - Kyiv City Heart Center, Kiev
  - Amosov National Institute of Cardiovascular Surgery, Kyiv

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Beeler R, Schoenenberger AW, Bauer P, Kobza R, Bergner M, Mueller X, Schlaepfer R, Zuber M, Erne S, Erne P. Improvement of cardiac function with device-based diaphragmatic stimulation in chronic heart failure patients: the randomized, open-label, crossover Epiphrenic II Pilot Trial. Eur J Heart Fail. 2014 Mar;16(3):342-9. doi: 10.1002/ejhf.20. Epub 2013 Dec 6. PMID 24464736
- [Result] Roos M, Kobza R, Jamshidi P, Bauer P, Resink T, Schlaepfer R, Stulz P, Zuber M, Erne P. Improved cardiac performance through pacing-induced diaphragmatic stimulation: a novel electrophysiological approach in heart failure management? Europace. 2009 Feb;11(2):191-9. doi: 10.1093/europace/eun377. PMID 19168496
- [Result] Jorbenadze A, Shaburishvili N, Mirro M, Zuber M, Erne P, Shaburishvili T. First-In-Human Visone Heart Failure Study: Asymptomatic Diaphragmatic Stimulation For Chronic Heart Failure With Reduced Ejection Fraction: Case Report. Journal of the American College of Cardiology. 2020;75(11) Supplement 1
- See also: Proof of concept therapeutic feasibility study of chronic ADS in post CABG heart failure patients — https://clinicaltrials.gov/ct2/show/NCT00769678